CLINICAL TRIAL: NCT03444129
Title: Pilot Evaluation of an Interactive Health Game Designed to Promote Healthy Eating and Physical Activity on Older Adults.
Brief Title: Pilot Evaluation of an Interactive Health Game
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Amparo Castillo, Training and Research Coordinator, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016-0218; 5P30AG022849 (NIH)
Record Dates: First submitted 2017-11-15; First posted 2018-02-23 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2018-02

CONDITIONS: Health Behavior; Health Attitude
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): This group will participate in a health education workshop with weekly sessions (control group)
  Interventions: Behavioral: Healthy eating workshop
- Game (Experimental): This group will participate in the health education workshop plus the interactive health game (intervention group).
  Interventions: Behavioral: Healthy eating workshop and interactive health game

INTERVENTIONS:
Behavioral: Healthy eating workshop and interactive health game — The intervention sessions will be weekly for 6 weeks and will involve participation in health education workshop and interactive health game. Sessions may last up to 2 hours and will be held at designated times/days at a Chicago Church.
  Arms: Game
Behavioral: Healthy eating workshop — The intervention sessions will be weekly for 6 weeks and will involve participation in health education workshop. Sessions may last up to 2 hours and will be held at designated times/days at a Chicago Church.
  Arms: Control

SUMMARY:
Broad, diverse, and innovative efforts are needed to address the growing dual public health challenges of obesity and diabetes, especially for those at increased risk like minority older adults. The emerging field of health games offers an innovative opportunity to reach populations to provide healthy eating and physical activity messages. Little research has focused on the use of health games specifically tailored for older adults. This study builds upon a health game designed to provide knowledge, facilitate movement, enhance motivation, and encourage healthy eating (HE) and physical activity (PA) behaviors in youth. This study will adapt, implement, and evaluate the feasibility, acceptability, adherence, and preliminary outcomes of the game among overweight/obese African American older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 65 years
* Overweight or obese (25kg/m2 ≤ BMI < 40kg/m2)
* African American/Black by self-report
* Risk factors for diabetes (based on adapted ADA risk test)

Exclusion Criteria:

* Adults with cognitive impairments, based on the adapted Mental Status Questionnaire (MSQ).
* Health conditions that preclude participation in physical activity program, based on the Exercise Assessment and Screener for You (EASY) physical activity screener.
* Already diagnosed with diabetes by self-report
* Currently engaging in vigorous physical activity
* Non-English speaking
* Does not meet inclusion criteria

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2018-03-10 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Eating habits | 6 weeks
  Eating habits will be assessed using the Visually-Enhanced Food Behavior Checklist.
Physical activity patterns | 6 weeks
  Physical activity patterns will be assessed using the short version of the International Physical Activity Questionnaire (IPAQ).
Motivation | 6 weeks
  Behavioral motivation questions will include Stage of change and confidence items to assess motivation (i.e., readiness) or achievement of behavioral goals.

SECONDARY OUTCOMES:
Weight | 6 weeks
  Weight will be measured using a digital scale
Adherence | 6 weeks
  Adherence will be measured by a count of the sessions attended.
Short International Physical Activity Questionnaire | 6 weeks
  Acceptability will be measured using this survey
MPP Acceptability Survey | 6 weeks
  This survey is about the participants experiences using MyPlatePicks (MPP) game
MPP stages of change survey | 6 week s
  acceptability will be measured using this survey

CONTACTS AND LOCATIONS:
Overall Officials: Amparo Castillo, PhD, Principal Investigator — UIC; Laurie Ruggiero, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No